CLINICAL TRIAL: NCT02911792
Title: Effect of Farxiga on Renal Function and Size in Type 2 Diabetic Patients With Hyperfiltration
Acronym: Hyper
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160262H
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperfiltering; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin; Glipizide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dapagliflozin/Hyperfiltration (Experimental): Subjects with eGFR above 125 ml/min per 1.73 m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization will have Dapagliflozin added to current metformin.
  Interventions: Drug: Dapagliflozin
- Metformin/Hyperfiltration (Active Comparator): Subjects who Drug naïve we will give Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization will have Metformin- XR, 1000 mg/day added. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Interventions: Drug: Metformin; Drug: Glipizide 5 MG
- Dapagliflozin/Normofiltration (Experimental): Subjects with eGFR below 124 ml/min per 1.73 m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization will have add Dapagliflozin added to current metformin.
  Interventions: Drug: Dapagliflozin
- Metformin/Normofiltration (Active Comparator): Subjects with eGFR below 124 ml/min per 1.73m2 drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Interventions: Drug: Metformin; Drug: Glipizide 5 MG

INTERVENTIONS:
Drug: Dapagliflozin — SGLT2 inhibitor
  Other Names: Farxiga
  Arms: Dapagliflozin/Hyperfiltration; Dapagliflozin/Normofiltration
Drug: Metformin — Oral diabetes medicine that helps control blood sugar levels.
  Other Names: Metformin-XR
  Arms: Metformin/Hyperfiltration; Metformin/Normofiltration
Drug: Glipizide 5 MG — Oral diabetes medicine that helps control blood sugar levels.
  Arms: Metformin/Hyperfiltration; Metformin/Normofiltration

SUMMARY:
The investigators propose to treat newly diagnosed, hyperfiltering T2DM patients with or without microalbuminuria with dapagliflozin or metformin for 4 months. The metformin-treated group will serve as controls for improved glycemic control, since the investigators have shown that insulin therapy to normalize A1c reduces hyperfiltration and kidney size in T1DM patients.

DETAILED DESCRIPTION:
Hyperfiltration is a characteristic feature in experimental models of diabetes and is causally related to an increase in intraglomerular pressure. In newly diagnosed diabetic patients, both type 1 and type 2, hyperfiltration and enlarged kidney size commonly are observed, and these hemodynamic/anatomic abnormalities are associated with an increased risk for the development of diabetic nephropathy.

In poorly controlled diabetic individuals, the filtered load of glucose is markedly increased and glucose - with sodium - reabsorption by the SGLT2 transporter in the proximal tubule is augmented. As a consequence sodium delivery to the macula densa is reduced, making the kidney think that it is under perfused and this results in afferent renal arteriolar vasodilation. The efferent arteriole of the hyperfiltrating diabetic kidney also is hypersensitive to angiotensin II despite the absence of systemic RAS activation. The net result of these hemodynamic changes is an increase in intraglomerular pressure and hyperfiltration. Further, angiotensin is a potent growth factor and contributes to the increase in size of individual glomeruli and total kidney size. Since the intraglomerular pressure is related to the radius (r3) by the Law of LaPlace, the increase in glomerular size also contributes to hyperfiltration.

Based upon the preceding sequence, it follows that a drug that blocks glucose, along with sodium, reabsorption in the proximal tubule would enhance sodium delivery to the macula densa, cause afferent renal arteriolar constriction, reduce intraglomerular pressure/hyperfiltration, and decrease kidney size. In hyperfiltering diabetic patients with microalbuminuria, the investigators also would expect the microalbuminuria to decrease. Consistent with this scenario, animal studies have documented that both acute and chronic inhibition of SGLT2 decreases hyperfiltration and prevents diabetic nephropathy. A recent study in hyperfiltering type 1 diabetic patients treated with empagliflozin has provided additional support for the tubular glomerular feedback hypothesis.

The investigators propose to treat newly diagnosed, hyperfiltering T2DM patients with or without microalbuminuria with dapagliflozin or metformin for 4 months. The metformin-treated group will serve as controls for improved glycemic control, since the investigators have shown that insulin therapy to normalize A1c reduces hyperfiltration and kidney size in T1DM patients

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, drug naïve, hyperfiltering and normofiltration patients with type 2 diabetes mellitus (T2DM)
* Hyperfiltration is defined by GFR >135 ml/min•1.73m2
* Normofiltration by a GFR = 90-134 ml/min•1.73m2
* BMI = 20-45 kg/m2
* HbA1c = 7.5% to 12%
* Willingness to participate in the 16 week study protocol
* Hematocrit >34% --BP < 145/90 mmHg

Exclusion Criteria:

* > 300 mg/day albumin excretion
* Ingestion of medications known to interfere with the renin-angiotensin system or renal function, including diuretic therapy
* Hospitalization for unstable angina, history of recent macrovascular (MI/stroke/TIA/ACS) disease, coronary artery revascularization (within 2 months prior to enrollment)
* Proliferative diabetic retinopathy
* History of cancer or major organ system disease
* New York Heart class II-IV heart failure Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3x ULN or total bilirubin > 2.0 mg/dL (34.2 µmo/L)
* Treatment with steroids, beta blockers, alpha blockers, antiobesity drugs
* Pregnant or nursing mothers
* Premenopausal females who are not practicing acceptable contraceptive methods Participation in another trial with an investigational drug within 30 days Alcohol or drug abuse within the preceding 6 months
* Any condition, psychiatric or medical, which in the opinion of the investigator would interfere with the successful completion of the study
* Orthostatic hypotension (> 15/10 mmHg decrease upon standing for 3 minutes)
* Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen, Hepatitis C virus antibody and HIV
* Volume depleted patients
* Estimated glomerular filtration rate <60 mL/min•1.73m2. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University Health Systems Texas Diabetic Institute, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available

REFERENCES:
- [Background] Hostetter TH, Troy JL, Brenner BM. Glomerular hemodynamics in experimental diabetes mellitus. Kidney Int. 1981 Mar;19(3):410-5. doi: 10.1038/ki.1981.33. PMID 7241881
- [Background] Brenner BM, Hostetter TH, Olson JL, Rennke HG, Venkatachalam MA. The role of glomerular hyperfiltration in the initiation and progression of diabetic nephropathy. Acta Endocrinol Suppl (Copenh). 1981;242:7-10. No abstract available. PMID 6940408
- [Background] Hostetter TH, Rennke HG, Brenner BM. The case for intrarenal hypertension in the initiation and progression of diabetic and other glomerulopathies. Am J Med. 1982 Mar;72(3):375-80. doi: 10.1016/0002-9343(82)90490-9. No abstract available. PMID 7036732
- [Background] Ruggenenti P, Porrini EL, Gaspari F, Motterlini N, Cannata A, Carrara F, Cella C, Ferrari S, Stucchi N, Parvanova A, Iliev I, Dodesini AR, Trevisan R, Bossi A, Zaletel J, Remuzzi G; GFR Study Investigators. Glomerular hyperfiltration and renal disease progression in type 2 diabetes. Diabetes Care. 2012 Oct;35(10):2061-8. doi: 10.2337/dc11-2189. Epub 2012 Jul 6. PMID 22773704
- [Background] Jerums G, Premaratne E, Panagiotopoulos S, MacIsaac RJ. The clinical significance of hyperfiltration in diabetes. Diabetologia. 2010 Oct;53(10):2093-104. doi: 10.1007/s00125-010-1794-9. Epub 2010 May 23. PMID 20496053
- [Background] Magee GM, Bilous RW, Cardwell CR, Hunter SJ, Kee F, Fogarty DG. Is hyperfiltration associated with the future risk of developing diabetic nephropathy? A meta-analysis. Diabetologia. 2009 Apr;52(4):691-7. doi: 10.1007/s00125-009-1268-0. Epub 2009 Feb 7. PMID 19198800
- [Background] Tuttle KR, Bruton JL, Perusek MC, Lancaster JL, Kopp DT, DeFronzo RA. Effect of strict glycemic control on renal hemodynamic response to amino acids and renal enlargement in insulin-dependent diabetes mellitus. N Engl J Med. 1991 Jun 6;324(23):1626-32. doi: 10.1056/NEJM199106063242304. PMID 2030719
- [Background] Stanton RC. Sodium glucose transport 2 (SGLT2) inhibition decreases glomerular hyperfiltration: is there a role for SGLT2 inhibitors in diabetic kidney disease? Circulation. 2014 Feb 4;129(5):542-4. doi: 10.1161/CIRCULATIONAHA.113.007071. Epub 2013 Dec 13. No abstract available. PMID 24334174
- [Background] Abdul-Ghani MA, Norton L, Defronzo RA. Role of sodium-glucose cotransporter 2 (SGLT 2) inhibitors in the treatment of type 2 diabetes. Endocr Rev. 2011 Aug;32(4):515-31. doi: 10.1210/er.2010-0029. Epub 2011 May 23. PMID 21606218
- [Background] Vallon V, Richter K, Blantz RC, Thomson S, Osswald H. Glomerular hyperfiltration in experimental diabetes mellitus: potential role of tubular reabsorption. J Am Soc Nephrol. 1999 Dec;10(12):2569-76. doi: 10.1681/ASN.V10122569. PMID 10589696
- [Background] Cherney DZ, Perkins BA, Soleymanlou N, Maione M, Lai V, Lee A, Fagan NM, Woerle HJ, Johansen OE, Broedl UC, von Eynatten M. Renal hemodynamic effect of sodium-glucose cotransporter 2 inhibition in patients with type 1 diabetes mellitus. Circulation. 2014 Feb 4;129(5):587-97. doi: 10.1161/CIRCULATIONAHA.113.005081. Epub 2013 Dec 13. PMID 24334175
- [Background] Zatz R, Dunn BR, Meyer TW, Anderson S, Rennke HG, Brenner BM. Prevention of diabetic glomerulopathy by pharmacological amelioration of glomerular capillary hypertension. J Clin Invest. 1986 Jun;77(6):1925-30. doi: 10.1172/JCI112521. PMID 3011862
- [Background] Taal MW, Brenner BM. Renoprotective benefits of RAS inhibition: from ACEI to angiotensin II antagonists. Kidney Int. 2000 May;57(5):1803-17. doi: 10.1046/j.1523-1755.2000.00031.x. PMID 10792600
- [Background] Anderson S, Vora JP. Current concepts of renal hemodynamics in diabetes. J Diabetes Complications. 1995 Oct-Dec;9(4):304-7. doi: 10.1016/1056-8727(95)80028-d. PMID 8573753
- [Background] Ellis EN, Steffes MW, Goetz FC, Sutherland DE, Mauer SM. Glomerular filtration surface in type I diabetes mellitus. Kidney Int. 1986 Apr;29(4):889-94. doi: 10.1038/ki.1986.82. PMID 3712971
- [Background] Schwieger J, Fine LG. Renal hypertrophy, growth factors, and nephropathy in diabetes mellitus. Semin Nephrol. 1990 May;10(3):242-53. PMID 2190281
- [Background] Malatiali S, Francis I, Barac-Nieto M. Phlorizin prevents glomerular hyperfiltration but not hypertrophy in diabetic rats. Exp Diabetes Res. 2008;2008:305403. doi: 10.1155/2008/305403. PMID 18769499
- [Background] Thomson SC, Rieg T, Miracle C, Mansoury H, Whaley J, Vallon V, Singh P. Acute and chronic effects of SGLT2 blockade on glomerular and tubular function in the early diabetic rat. Am J Physiol Regul Integr Comp Physiol. 2012 Jan 1;302(1):R75-83. doi: 10.1152/ajpregu.00357.2011. Epub 2011 Sep 21. PMID 21940401
- [Background] Pei F, Li BY, Zhang Z, Yu F, Li XL, Lu WD, Cai Q, Gao HQ, Shen L. Beneficial effects of phlorizin on diabetic nephropathy in diabetic db/db mice. J Diabetes Complications. 2014 Sep-Oct;28(5):596-603. doi: 10.1016/j.jdiacomp.2014.04.010. Epub 2014 Apr 24. PMID 24927646
- [Background] Bakker J, Olree M, Kaatee R, de Lange EE, Moons KG, Beutler JJ, Beek FJ. Renal volume measurements: accuracy and repeatability of US compared with that of MR imaging. Radiology. 1999 Jun;211(3):623-8. doi: 10.1148/radiology.211.3.r99jn19623. PMID 10352583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Type 2 Diabetes patients recently diagnosed either drug naive or or metformin in good general health with eGFR either above 125 or below 124 ml/min per 1.73 m2 were recruited
Pre-assignment Details: eGFR Above 125 ml/min per 1.73m2 included in the HYPERFILTRATION GROUPS.
  eGFR Below 124 ml/min per 1.73m2 included in the NORMOFILTRATION GROUPS
Groups:
- Dapagliflozin/Hyperfiltration: Subjects with eGFR equal or above 125 ml/min/1.73m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization we will add Dapagliflozin to current metformin.
  Dapagliflozin: SGLT2 inhibitor
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
- Metformin?Hyperfiltration: Subjects eGFR equal or above 125 ml/min/1.73m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
- Dapagliflozin/Normofiltration: Subjects eGFR equal or below 124 ml/min/1.73m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization we will add Dapagliflozin to current metformin.
  Dapagliflozin: SGLT2 inhibitor
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
- Metformin/Normofiltration: Subjects with eGFR equal or below 125 ml/min/1.73m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
Period: Overall Study
Arm/Group | Dapagliflozin/Hyperfiltration | Metformin?Hyperfiltration | Dapagliflozin/Normofiltration | Metformin/Normofiltration
Started | 18 | 18 | 18 | 18
Completed | 15 | 15 | 15 | 15
Not Completed | 3 | 3 | 3 | 3
Not completed — Lost to Follow-up | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Type 2 diabetes in good general health with eGFR above and below 125 ml/min per 1.73m2 who are either drug naive or taking metformin.
Groups:
- Dapagliflozin/Hyperfiltration: Subjects with eGFR above 125 ml/min per 1.73 m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization we will add Dapagliflozin to current metformin.
  Dapagliflozin: SGLT2 inhibitor
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
- Metformin/Hyperfiltration: Subjects with GFR above 125 ml/min per 1.73m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
- Dapagliflozin/Normofiltration: Subjects with eGFR below 124 ml/min per 1.73 m2 will be randomized to dapagliflozin, 5 mg/day. After 2 weeks (Visit 5), dapagliflozin will be increased to 10 mg/day, Subjects who are taking Metformin at time of randomization we will add Dapagliflozin to current metformin.
  Dapagliflozin: SGLT2 inhibitor
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
- Metformin/Normofiltration: Subjects with GFR below 124 ml/min per 1.73m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin/Hyperfiltration | Metformin/Hyperfiltration | Dapagliflozin/Normofiltration | Metformin/Normofiltration | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (5) | 55 (5) | 51 (6) | 54 (4) | 52 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 8 | 9 | 36
  Male | 6 | 5 | 7 | 6 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: GFR (Glomerular Filtration Rate) Change After Treatment
Description: Change from baseline in GFR after treatment from baseline to 4 months
Time Frame: 4 months
Population: Type 2 diabetes in good general health with eGFR above or below125 ml/min/1.73m^2 either drug naïve or on metformin.
Measure: Mean (Standard Error); unit: ml/min/1.73m^2
Groups:
- Metformin/Hyperfiltration: Subjects with eGFR above 125 ml/min per 1.73m2 drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
Arm/Group | Dapagliflozin/Hyperfiltration | Metformin/Hyperfiltration | Dapagliflozin/Normofiltration | Metformin/Normofiltration
Number analyzed (Participants) | 15 | 15 | 15 | 15
ml/min/1.73m^2 | 22 (6) | 1 (5) | 8 (3) | 0 (4)

ADVERSE EVENTS:
Time Frame: All adverse events were recorded during the entire 4 months period of the study
Description: Adverse events collection relied on volunteers reports and physical examination with periodic laboratory analysis, as necessary
Groups:
- Metformin/Hyperfiltration: Subjects with eGFR above 125 ml/min per 1.73 m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
- Metformin/Normofiltration: ubjects with eGFR below 124 ml/min per 1.73 m2 who are drug naïve will receive Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).Subject who are on metformin at time of randomization we will add Glipizide 5 mg( to be increased to 10 mg at Visit 5), Subject who are on Glipizide at time of randomization we will add Metformin- XR, 1000 mg/day. After 2 weeks (Visit 5), metformin will be increased to 1000 mg bid (twice a day).
  Metformin: Oral diabetes medicine that helps control blood sugar levels.
  Glipizide 5 MG: Oral diabetes medicine that helps control blood sugar levels.
Arm/Group | Dapagliflozin/Hyperfiltration | Metformin/Hyperfiltration | Dapagliflozin/Normofiltration | Metformin/Normofiltration
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 3/15 | 4/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin/Hyperfiltration (N=15) | Metformin/Hyperfiltration (N=15) | Dapagliflozin/Normofiltration (N=15) | Metformin/Normofiltration (N=15)
Genital Mycotic Infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Mild Hypoglycemia (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT02911792/Prot_SAP_000.pdf